CLINICAL TRIAL: NCT06370884
Title: An Open-Label, Pilot Clinical Trial To Test The Safety And Feasibility Of Intestinal Microbiota Transplantation In Patients Undergoing Colon Resection
Brief Title: Intestinal Microbiota Transplantation in Patients Undergoing Colon Resection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SURG-2023-29833
Record Dates: First submitted 2024-03-04; First posted 2024-04-17 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Clostridioides Difficile Infection; Colonic Surgery
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: This is a phase 1 pilot clinical trial that will evaluate the initial safety and feasibility of intestinal microbiota transplantation (IMT) in patients undergoing colon resection.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMT group (Experimental): individuals of the ages of 18-75 with a history of diverticulitis or sigmoid colon cancer will be enrolled to have a feeding tube placed at the time of surgery and receive either IMT solution
  Interventions: Drug: IMT

INTERVENTIONS:
Drug: IMT — a feeding tube placed at the time of surgery and receive IMT solution on postoperative day 2-3 (at least 48 hours following IV antibiotics) with the subsequent removal of the feeding tube.

SUMMARY:
This is a single-center, open-label study for safety and feasibility of IMT in patients undergoing colonic surgery. After consent, individuals of the ages of 18-75 with a history of diverticulitis or sigmoid colon cancer will be enrolled to have a feeding tube placed at the time of surgery and receive IMT solution on postoperative day 2-3 (at least 48 hours following IV antibiotics) with the subsequent removal of the feeding tube. Prior to administration of IMT, recipients will be screened for inclusion/exclusion criteria, interviewed for medical history and medications, and consented. Additionally, prior to undergoing IMT, baseline blood and fecal samples will be collected. The use of a nasogastric feeding tube has specifically been chosen over colonoscopic introduction of the IMT. This is because colonoscopy introduces increased intraluminal carbon dioxide and pressure as well as mechanical stress on the colon in the setting of a newly created bowel anastomosis, which may contribute to the potential risk of anastomotic disruption. The nasogastric feeding tube will be placed while the patient is under anesthesia under direct visualization to minimize any risk of bowel perforation, albeit very low. The study will specifically utilize a 10F 43" Corpak feeding tube (Halyard Health, Alpharetta, GA). Patients will be monitored while in-patient in person. Following discharge, they will undergo follow-up either by phone, video or in-person visit, or via online survey of symptoms and chronic medical conditions potentially related to IMT, beginning on the day following discharge through post-operative day 14, and then monthly up to 6 months post- IMT to screen for SAEs and AEs. Screening for SAEs and AEs will be done using a symptom questionnaire as well as by asking patients during our interview. Fecal samples will be collected from participants on months one, three and six post-IMT to assess for changes in recipient microbiome (engraftment kinetics).

ELIGIBILITY:
Inclusion Criteria:

* Able/willing to provide informed consent
* Between 18-75 years of age
* Undergoing surgery for a history of diverticulitis or sigmoid colon cancer.
* Able to provide fecal samples
* Stated willingness to comply with all study procedures and availability for the duration of trial to follow-up by telephone, in-person, email, and/or video visits or correspondence

Exclusion Criteria:

* Any history of inflammatory bowel disease
* Pregnancy or breastfeeding. A pregnancy test will be obtained from females of child- bearing potential on the proposed day of IMT (prior to the receipt of IMT). Patients with a positive pregnancy test will be excluded. A negative result will be required for subjects who are females of child-bearing potential to receive IMT treatment.
* Life expectancy of < 6 months
* Presence of ileostomy or colostomy
* Known history of inflammatory bowel disease (Crohn's, Ulcerative Colitis)
* Patients on immunosuppressants (calcineurin inhibitors, prednisone ≥ 20 mg/day, methotrexate, azathioprine, immunosuppressive biologics, JAK inhibitors)
* Patients with neutropenia (an absolute neutrophil count < 0.5 x 109 cells/L) obtained on a complete blood count with differential at screening.
* History of solid organ or bone marrow transplant.
* Anticipated recurrent antibiotic use (e.g., patients with frequent urinary tract infections or sinusitis).
* History of severe anaphylactic food allergy.
* History of celiac disease.
* Patients receiving cancer chemotherapy, immunotherapy, or radiation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety of IMT in patients undergoing colon surgery | Day of surgery, post-op Day 1-14, Day30, Day60, Day90, Day120, Day150, Day180
  Collected via adverse event monitoring, to be reported as frequency, relatedness, expectedness, and severity of AEs/SAEs
compare fecal microbiota prior to and after IMT | Day -60-0, Day of surgery, post-op Day1-3, Day14, Day30, Day90, Day180
  Collected via stool sample collection, to be reported as sequenced microbial DNA profiles (alpha diversity, beta diversity)

SECONDARY OUTCOMES:
Evaluate engraftment of donor microbiota | Day -60-0, day of surgery, postoperative Day1-3, Day14
  ollected via stool sample, to be reported as sequenced microbial DNA profiles (alpha diversity, beta diversity). We will compare preoperative stool samples to samples collected post-transplant of the donor microbiota
Evaluate changes in circulating markers of inflammation: WBC | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported White blood count (WBC) is 10^9/liter, absolute number in 10^9, volume in liters
Evaluate changes in circulating markers of inflammation: Hemoglobin | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Hemoglobin is grams/deciliter (g/dL), weight in grams, volume in deciliters
Evaluate changes in circulating markers of inflammation: Platelets | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Platelets is 10^9/liter, absolute number in 10^9, volume in liters
Evaluate changes in circulating markers of inflammation: Electrolytes | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Sodium, potassium, chloride, carbon dioxide are millimole/liter (mmol/L), amount of substance in millimoles, volume in liters
Evaluate changes in circulating markers of inflammation | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Blood urea nitrogen, creatinine, glucose, magnesium, total bilirubin, prealbumin are milligrams/deciliter (mg/dL) weight in milligrams, volume in deciliters
Evaluate changes in circulating markers of inflammation: alkaline phosphatase | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine transaminase (ALT) are units/liter (U/L) amount of substance in Units, volume in liters
Evaluate changes in circulating markers: Albumin | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Total protein, albumin are grams/liter (g/L) weight in grams, volume in liters
Evaluate changes in microbial metabolites: Fecal short-chain fatty-acids | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Fecal short-chain fatty acids are millimole/kilogram (mmol/kg) amount of substance in millimoles, weight in kilograms
Evaluate changes in microbial metabolites: Fecal IgA | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via blood sample with standard laboratory values reported Fecal IgA is nanograms IgA/ milligram of stool (ng IgA/mg stool) weight of IgA in nanograms, weight of stool in milligrams
Compare baseline microbiome characteristics with changes over time after IMT | Day -60-0, day of surgery, postoperative Day1-3, Day14, Day30, Day90, Day180
  Collected via stool sample, to be reported as sequenced microbial DNA profiles (alpha diversity, beta diversity). We will compare preoperative stool samples to samples collected post-transplant of the donor microbiota across all time points.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Jahansouz, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States